CLINICAL TRIAL: NCT06799195
Title: A Phase II Randomized Trial to Optimize GVHD Prophylaxis After Allogeneic Hematopoietic Cell Transplantation in Older Adults With Hematological Malignancies: the PROMISE Trial
Brief Title: Optimizing GVHD Prophylaxis After Allogeneic Hematopoietic Cell Transplantation
Acronym: PTCYGVHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0094-25-FB
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Hematological Malignancies; Graft-versus-Host Disease (GVHD)
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; GVHD Prophylaxis; Sirolimus; Mycophenolate Mofetil (MMF); Health-Related Quality of Life (HRQoL); Randomized Controlled Trial
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease | interventions — Cyclophosphamide; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, phase II trial comparing two graft-versus-host disease (GVHD) prophylaxis regimens in older adults undergoing allogeneic hematopoietic stem cell transplantation. Participants are randomized into two arms: high-dose (standard care) versus attenuated-dose post-transplant cyclophosphamide (PTCy), both in addition to sirolimus and mycophenolate mofetil (MMF).
Masking Description: Not applicable; the study is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attenuated-dose post-transplant cyclophosphamide (PTCy) Arm (Experimental): Participants will receive attenuated-dose post-transplant cyclophosphamide (PTCy) at 25 mg/kg on days +3 and +4 after allogeneic hematopoietic stem cell transplantation. This is in addition to sirolimus and mycophenolate mofetil (MMF) for graft-versus-host disease (GVHD) prophylaxis.
  Interventions: Drug: Attenuated-dose Cyclophosphamide; Drug: Sirolimus; Drug: Mycophenolate Mofetil (MMF)
- High-dose post-transplant cyclophosphamide (PTCy) Arm: Standard of Care (Active Comparator): Participants will receive high-dose post-transplant cyclophosphamide (PTCy) at 50 mg/kg on days +3 and +4 after allogeneic hematopoietic stem cell transplantation. This is in addition to sirolimus and mycophenolate mofetil (MMF) for GVHD prophylaxis.
  Interventions: Drug: High-dose Cyclophosphamide; Drug: Sirolimus; Drug: Mycophenolate Mofetil (MMF)

INTERVENTIONS:
Drug: Attenuated-dose Cyclophosphamide — Cyclophosphamide administered at an attenuated dose of 25 mg/kg on days +3 and +4 post-transplant for GVHD prophylaxis.
  Arms: Attenuated-dose post-transplant cyclophosphamide (PTCy) Arm
Drug: High-dose Cyclophosphamide — Cyclophosphamide administered at the standard high dose of 50 mg/kg on days +3 and +4 post-transplant for GVHD prophylaxis.
  Arms: High-dose post-transplant cyclophosphamide (PTCy) Arm: Standard of Care
Drug: Sirolimus — Sirolimus is started on day +5 with a loading dose of 6 mg, followed by a maintenance dose of 2 mg daily, adjusted to target trough levels of 8-12 ng/mL. Sirolimus taper is recommended to start at day +90 and to be completed by day +180, provided there is no evidence of acute GVHD.
Drug: Mycophenolate Mofetil (MMF) — MMF is started on day +5 at a dose of 15 mg/kg per dose (maximum 1 g per dose) three times daily. MMF is generally discontinued by day +35 in the absence of GVHD.

SUMMARY:
This study will compare post-transplant health-related quality of life following the use of standard versus attenuated dose of post-transplant cyclophosphamide in addition to two-drug graft-versus-host disease (GVHD) prophylaxis among recipients of allogeneic hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
This is a single-center phase II study of 126 participants (63 per arm) with hematological malignancies. Participants will be randomized to receive high doses (standard arm) or attenuated doses of cyclophosphamide in addition to two-drug GVHD prophylaxis. Participants will be monitored for health-related quality of life [Functional Assessment of Cancer Therapy-Bone Marrow Transplant, FACT-BMT(1)], functional outcomes (Karnofsky Performance Scale (KPS), activities of daily living, instrumental activities of daily living, Clock-in-the-Box Test, Fried Frailty Index, fall history, BMI, and Geriatric Depression Scale-15, GVHD, relapse, survival, and toxicities (using Common Terminology Criteria for Adverse Events, CTCAE version 5.0).

ELIGIBILITY:
Inclusion criteria:

* Adults aged 60 years or older
* Diagnosis of a hematological malignancy or other serious hematological disorder that requires an allogeneic hematopoietic cell transplantation
* Planned to receive any reduced-intensity conditioning regimen (any graft source is acceptable) and availability of human leukocyte antigen (HLA)-matched donor at HLA loci A, B, C, and HLA-DR beta chain antigen (DRB1)
* Karnofsky Performance Status (KPS) of 70% or higher.

Exclusion criteria:

* Previous history of one or more prior allogeneic stem cell transplants (i.e., second or third allogeneic transplant)
* Planned use of high doses of cyclophosphamide (e.g., a total cyclophosphamide dose of approximately 50 mg/kg or more) as part of the conditioning regimen prior to allogeneic stem cell transplant. A lower dose of cyclophosphamide (e.g., fludarabine, cyclophosphamide, and low-dose total body irradiation regimen that uses 2 doses of cyclophosphamide at 14.5 mg/kg) is acceptable.
* Known diagnosis of liver cirrhosis or other advanced liver disease that may impact cyclophosphamide metabolism.
* Diagnosis of myelofibrosis
* Creatinine clearance less than 40 mL/min/1.73 m², which may increase the risk of hemorrhagic cystitis with post-transplant cyclophosphamide (PTCy)
* Systolic cardiac dysfunction with an ejection fraction of less than 45%.
* Use of a haploidentical or mismatched donor.
* Any other condition judged by the physician to increase the risk of toxicities associated with PTCy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life as Measured by Functional Assessment of Cancer Therapy-Bone Marrow Transplantation | Baseline and 3 months post-transplant
  The health-related quality of life will be assessed using the Functional Assessment of Cancer Therapy-Bone Marrow Transplantation (FACT-BMT) trial outcome index (TOI). The FACT-BMT is a validated, patient-reported questionnaire that measures physical and functional well-being specifically in bone marrow transplant recipients. Higher scores indicate better quality of life. The primary outcome is to compare the FACT-BMT TOI scores between the attenuated-dose PTCy arm and the high-dose PTCy arm at 3 months post-transplant.

SECONDARY OUTCOMES:
Change in Karnofsky Performance Scale | Baseline and 3 months post-transplant
  Karnofsky Performance Scale (KPS) is a validated tool ranging from 0 (death) to 100 (normal activity). Higher scores indicate better functional status.
Change in Activities of Daily Living | Baseline and 3 months post-transplant
  Activities of Daily Living (ADL) measures basic self-care tasks such as bathing and dressing. The typical total score ranges from 0 to 6, with higher scores indicating better functional status.
Change in Instrumental Activities of Daily Living | Baseline and 3 months post-transplant
  Change in Instrumental Activities of Daily Living (IADL) assesses more complex tasks (e.g., handling finances). Total scores typically range from 0 to 8 or 0 to 14 (depending on the version), with higher scores indicating greater independence.
Change in Fried Frailty Index | Baseline and 3 months post-transplant
  The Fried Frailty Index assesses five components (weight loss, exhaustion, grip strength, walking speed, and physical activity). A higher total score indicates greater frailty.
Change in Clock-in-the-Box Test | Baseline and 3 months post-transplant
  This is a brief test of visuospatial and executive function, typically scored on accuracy of clock drawing/placement (range 0-8). Higher scores suggest better cognitive performance.
Change in History of Falls | Baseline and 3 months post-transplant
  The number of falls, if any, will be collected since baseline. Results will be analyzed as the proportion of participants experiencing ≥1 fall over the time frame, or as the difference in mean (or median) number of falls between arms.
Change in Body Mass Index | Baseline and 3 months post-transplant
  Body Mass Index (BMI) is calculated as weight (kg) / [height (m)]² (kg/m²). Higher or lower values do not necessarily indicate "better" or "worse" status by themselves but will be compared between arms for changes from baseline.
Change in Geriatric Depression Scale-15 | Baseline and 3 months post-transplant
  The Geriatric Depression Scale-15 (GDS-15) is a 15-item screening tool for depression in older adults (scores 0-15). Higher scores indicate more severe depression.
Gaft-Versus-Host Disease-Free, Relapse-Free Survival | From date of transplant to 1 year post-transplant
  Graft-Versus-Host Disease (GRFS) is defined as the time from transplant to the first occurrence of grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, disease relapse or progression, or death from any cause. An event is counted when any of these conditions are met. The GRFS at 1 year post-transplant will be compared between the two treatment arms.
Overall Survival at 1 Year Post-Transplant and Event-Free Survival | From date of transplant to 1 year post-transplant
  Overall Survival (OS) is defined as survival from the date of transplant until death from any cause. Event-Free Survival (EFS) is defined as survival from the date of transplant without disease relapse or progression. The study will compare the proportion of participants alive (for OS) and without relapse or progression (for EFS) at 1 year post-transplant between the two treatment arms
Cumulative Incidence of Transplant-Related Mortality | From date of transplant to 1 year post-transplant
  Transplant-related mortality (TRM) is defined as death from causes other than disease relapse or progression. The study will estimate and compare the cumulative incidence of TRM at 1 year post-transplant between the two treatment arms.
Cumulative Incidence of Grade II-IV Acute GVHD | From date of transplant to 1 year post-transplant
  Acute graft-versus-host disease (GVHD) of grade II-IV is assessed using the Mount Sinai acute GVHD grading system. The study will estimate and compare the cumulative incidence of grade II-IV acute GVHD at 1 year post-transplant between the two treatment arms.
Cumulative Incidence of Chronic GVHD | From date of transplant to 1 year post-transplant
  Chronic GVHD is assessed using the NIH chronic GVHD grading system, which includes both classical chronic GVHD and overlap syndrome. The study will estimate and compare the cumulative incidence of chronic GVHD at 1 year post-transplant between the two treatment arms.
To determine the cumulative incidence and kinetics of hematologic recovery (neutrophil and platelet) among the two treatment arms | From date of transplant to day +28 and day +100 post-transplant
  Hematologic recovery is evaluated by time to neutrophil engraftment (absolute neutrophil count ≥ 500/mm³ for three consecutive days) and platelet engraftment (platelet count ≥ 20,000/mm³ or ≥ 50,000/mm³ without transfusion for seven days). The study will describe and compare the cumulative incidence and kinetics of neutrophil and platelet recovery by days +28 and +100 post-transplant between the two treatment arms.
Incidence of Grade III or Higher Adverse Events | From date of transplant to day +100 post-transplant
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The study will assess and compare the incidence of grade III or higher adverse events by day +100 post-transplant between the two treatment arms.
Cumulative Incidence of Grade II or Higher Infections | From date of transplant to 6 months post-transplant
  Infections will be graded according to Blood and Marrow Transplant Clinical Trials Network (BMT CTN) criteria. The study will estimate and compare the cumulative incidence of grade II or higher infections by 6 months post-transplant between the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Moataz Ellithi, MBChB, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luznik L, Pasquini MC, Logan B, Soiffer RJ, Wu J, Devine SM, Geller N, Giralt S, Heslop HE, Horowitz MM, Jones RJ, Litzow MR, Mendizabal A, Muffly L, Nemecek ER, O'Donnell L, O'Reilly RJ, Palencia R, Schetelig J, Shune L, Solomon SR, Vasu S, Ho VT, Perales MA. Randomized Phase III BMT CTN Trial of Calcineurin Inhibitor-Free Chronic Graft-Versus-Host Disease Interventions in Myeloablative Hematopoietic Cell Transplantation for Hematologic Malignancies. J Clin Oncol. 2022 Feb 1;40(4):356-368. doi: 10.1200/JCO.21.02293. Epub 2021 Dec 2. PMID 34855460
- [Background] Korngold R, Sprent J. Lethal graft-versus-host disease after bone marrow transplantation across minor histocompatibility barriers in mice. Prevention by removing mature T cells from marrow. J Exp Med. 1978 Dec 1;148(6):1687-98. doi: 10.1084/jem.148.6.1687. PMID 363972
- [Background] Wingard JR, Majhail NS, Brazauskas R, Wang Z, Sobocinski KA, Jacobsohn D, Sorror ML, Horowitz MM, Bolwell B, Rizzo JD, Socie G. Long-term survival and late deaths after allogeneic hematopoietic cell transplantation. J Clin Oncol. 2011 Jun 1;29(16):2230-9. doi: 10.1200/JCO.2010.33.7212. Epub 2011 Apr 4. PMID 21464398
- [Background] McQuellon RP, Russell GB, Cella DF, Craven BL, Brady M, Bonomi A, Hurd DD. Quality of life measurement in bone marrow transplantation: development of the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) scale. Bone Marrow Transplant. 1997 Feb;19(4):357-68. doi: 10.1038/sj.bmt.1700672. PMID 9051246